CLINICAL TRIAL: NCT02167932
Title: Impact of a Physical Activity Program on Biomarkers of Aging During Adjuvant or Neoadjuvant Chemotherapy for Breast Cancer
Brief Title: The Impact of a Physical Activity Program on Biomarkers of Aging During Chemotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1334
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer; Aging
Keywords: Breast Cancer; Walk With Ease; Physical Activity; Walking; Younger Women; Cancer; p16; Aging; Biomarkers; Biomarkers of Aging; Chemotherapy; Chemotherapy Treatment; Adjuvant Chemotherapy; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Neoplasms | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken collect p16 levels, CBC + Differential and senescence markers.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast Cancer Patients: Breast Cancer patients undergoing chemotherapy will participate in the Walk with Ease program during their treatment.
  Interventions: Behavioral: Walk With Ease

INTERVENTIONS:
Behavioral: Walk With Ease — Walk With Ease is the Arthritis Foundation's evidence-based walking intervention to help with fatigue and pain. The intervention is a self-directed program that helps guide participants in a safe and comfortable paced walking program with an ultimate goal of walking for 30 minutes a day, five days a week.
  Other Names: WWE

SUMMARY:
This study will look at whether or not participating in a physical activity intervention during chemotherapy for breast cancer can prevent a marker of aging called p16 from having a large increase after chemotherapy.

DETAILED DESCRIPTION:
Our research team has determined that p16INK4a - a biomarker of aging -- increases dramatically during chemotherapy and that p16 levels among patients of similar age are lower among those who exercise. We hypothesize that engagement in physical activity during chemotherapy will have a moderating effect on increases in p16 levels during chemotherapy. To test this hypothesis, we propose to enroll 48 patients age 21-64 with a Stage I-III breast cancer diagnosis who are about to start adjuvant or neoadjuvant chemotherapy in a physical activity intervention program. Our primary objective is to compare the change in p16 from baseline to end of chemotherapy for participants in this study (who are engaged in a physical activity intervention) to the mean change in p16 seen in a previous study of similar patients who did not participate in a physical activity intervention. As secondary objectives, we propose to evaluate (1) changes in treatment-related toxicity, physical function, fatigue, and quality of life between baseline, end of chemotherapy and 6 months post-chemotherapy, (2) the association of changes in p16 levels with changes in measures of treatment-related toxicity, physical function, fatigue, and quality of life, and (3) the association of changes in physical activity levels with changes in measures of treatment-related toxicity, physical function, fatigue, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 59 years of age, female (A similar trial LCCC 1226 explores physical activity in women 60 years and older and is now in progress.
* Histologically confirmed Stage I, II or III breast cancer (if the patient has had more than one breast cancer, then the most recent diagnosis)
* Scheduled to begin an appropriate adjuvant or neo-adjuvant chemotherapy regimen as defined by NCCN guidelines (www.nccn.org). Patients receiving anti-HER-2 therapy are eligible but the intervention will only be tested during the chemotherapy portion of the regimen.
* English speaking
* IRB approved, signed written informed consent
* Approval from their treating physician to engage in moderate-intensity physical activity
* Patient-assessed ability to walk and engage in moderate physical activity
* Willing and able to meet all study requirements.

Exclusion Criteria:

* One or more significant medical conditions that in the physician's judgment preclude participation in the walking or strength training intervention.
* Unable to walk or engage in moderate-intensity physical activity.

Ages: 21 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Breast Cancer Patients age 21-59
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2014-03; Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Compare the change in p16 from baseline to the end of chemotherapy for patients receiving a physical activity intervention to the historical value seen in a previous study | One Year
  Mean change in p16 levels measured between baseline to end of chemotherapy, as compared to the historical value seen in a previous study (LCCC810) of similar patients who did not participate in a physical activity intervention

SECONDARY OUTCOMES:
Measure the association of change in physical activity levels with change in with p16 levels from baseline to end of chemo and baseline to 6-months post. | One year
  Information obtained through patient-reported surveys and p16 levels obtained from blood samples between baseline to 6 month post-chemotherapy
Compare changes in p16 between patients who do and do not experience any grade 3/4 toxicities | One year
  Information obtained through physician and patient reported surveys.
Predict changes in physical function, fatigue, and quality of life over | One year
  This objective will use the surveys that measure physical function, fatigue and quality of life to see if they can make any predictions about how these domains may change over the course of chemotherapy.
Measure the association of change in physical activity levels with changes in physical function, fatigue, and quality of life measures | One year
  Changes will be measured over the course of the study
Measure the association of change in p16 levels with changes in physical function, fatigue, and quality of life measures | One year
  Changes will be measured over the course of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hyman B Muss, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Nyrop KA, Page A, Deal AM, Wagoner C, Kelly EA, Kimmick GG, Copeland A, Speca J, Wood WA, Muss HB. Association of self-directed walking with toxicity moderation during chemotherapy for the treatment of early breast cancer. Support Care Cancer. 2023 Dec 28;32(1):68. doi: 10.1007/s00520-023-08275-4. PMID 38153568
- See also: UNC Geriatric Oncology Program — https://unclineberger.org/patientcare/programs/geriatric